CLINICAL TRIAL: NCT04964115
Title: Post Acute Sequelae of SARS-CoV-2
Brief Title: Post Acute Sequelae of COVID-19
Acronym: PASC
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Carla Sevin, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 210436
Record Dates: First submitted 2021-05-13; First posted 2021-07-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Covid19; Sars-CoV-2 Infection; Dyspnea Caused by 2019-nCoV; COVID-19 Acute Respiratory Distress Syndrome; Pulmonary Fibrosis
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cohort study — This cohort study does not involve an intervention

SUMMARY:
COVID-19, a novel coronavirus, has caused widespread mortality and morbidity since it emerged in 2019. There is ongoing research and growing literature describing severe acute respiratory syndrome (SARS-COV-2). There is a growing population of individuals who have recovered from acute SARS-COV-2 infection. The long-term effects of COVID-19 are unknown. There are growing reports of sequelae after acute SARS-CoV-2 not limited to fatigue, dyspnea, reactive airway disease, organizing pneumonia, pulmonary fibrosis, pulmonary hypertension, pulmonary emboli, and tracheal disease. The incidence and natural history of these findings is unstudied.

DETAILED DESCRIPTION:
COVID-19 is a leading cause of death worldwide. The long-term effects of the virus are unknown. There is lack of reliable information about the natural history of post acute sequelae. Although there are limited evidence-based treatment guidelines, many patients receive unproven therapies. Given the mortality and morbidity associated with the illness and the growing number of patients who have survived COVID-19 the long-term effects are a growing area of inquiry. This study is designed to better understand the effects of SARS-CoV-2 that develop over time. This study will characterize the recovery process, epidemiology, and natural history of post-acute sequelae. This includes the clinical spectrum of recover and subsets of patients who have symptoms outside the standard course. Factors studied will include the individual, clinical context, severity of disease, duration of symptoms and the impact of treatment for acute SARS-CoV-2. This study will include a breadth of severity from those treated as outpatients, those requiring hospitalization, and those requiring critical care.

Key personnel will extract data recorded in the electronic health record (EHR) as part of routine clinical care in the evaluation in treatment of COVID-19 and its sequelae. Data such as incidence, prevalence, demographics, comorbidities, duration of illness, severity, level of medical care, measures of organ function, drug treatments, laboratory values, pulmonary function tests, computed tomography images, and other data from clinical care will be retrospectively entered into electronic data capture (REDCap).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* COVID-19 diagnosis
* Seen in a Vanderbilt clinic or affiliated health facility

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of COVID-19 seen at Vanderbilt or an affiliated health facility.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Natural history of recovery from COVID-19 | up to 5 years
  Incidence, prevalence, age, sex, BMI, presence of comorbid conditions (including diabetes, hypertension, immunosuppression, or chronic lung disease), duration of illness (in days), level of medical care (intensive care unit, inpatient or outpatient), drug therapies received, pulmonary function tests, and computed tomography images.

SECONDARY OUTCOMES:
Natural history of patients who do not recover from COVID-19 | up to 5 years
  Phenotypes of recovery (complete recovery, delayed recovery, no recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Carla M Sevin, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt_University MC, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No